CLINICAL TRIAL: NCT03934242
Title: Impact of Information Campaign's Alongside Maternity Staff About Bedding Infant
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19012
Record Dates: First submitted 2019-03-12; First posted 2019-05-01 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-04

CONDITIONS: Sudden Death in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New born group 1: New born who was born at the maternity of the CHU of Reims during a period of inclusion of one month, before nurses formation on the newborn's bedding
  Interventions: Other: Questionnaire on new born's bedding
- New born group 2: New born who was born at the maternity of the CHU of Reims during a period of inclusion of one month, after nurses formation on the newborn's bedding
  Interventions: Other: Questionnaire on new born's bedding

INTERVENTIONS:
Other: Questionnaire on new born's bedding — Questionnaire on new born's bedding (Child's position in the bed : dorsal, ventral or lateral, presence of pillow or stuffed in bed, presence of coverage and presence of the bed sharing) at two times (during hospitalisation and one month later)

SUMMARY:
It is now well established that infants should be placed on the back only in a SleepSack without coverage or plush or pillow on a firm mattress in a bedroom. Despite these old recommendations of good practice, deviations are observed and some infants are most always lying according to the recommended position. The goal is to assess the impact of an information campaign of staffs maternity of the CHU of Reims on the practices of the sleeping of infants to motherhood, and then at the home of the parents.

DETAILED DESCRIPTION:
Proposal for participation to the holders of parental authority of newborns eligible within 72 hours after the birth of the child. If acceptance of participation, the newborn will be included in the study. Participation in the study will not affect the medical care of the child. Participation in the study will consist of: a collection of data including the child sleeping mode, complete a questionnaire covering the child sleeping habits to motherhood and home during the 1st month of life. Information on the habits of sleeping in the home of the child will be collected via a phone call by an investigator. Inclusions will be held over 2 periods: one before and one after the completion of training of health care personnel regarding the sleeping of infants nursing staff training will consist of oral information by the investigative team and written information...

ELIGIBILITY:
Inclusion Criteria:

* born in reims CHU
* parents are 18 years old or more
* parents accept their participation in the study

Exclusion criteria :

* hospitalization in URIP / kangourou / neonatalogy
* needed baby warmer

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: every newborn
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
correct new born's bedding | Day 0
  Newborn's bedding will be considered correct if the newborn is lying alone (no bed sharing), in exclusive dorsal position (no ventral or lateral position), in a bed without pillow, without blanket and without soft toy.
correct new born's bedding | month 1
  Newborn's bedding will be considered correct if the newborn is lying alone (no bed sharing), in exclusive dorsal position (no ventral or lateral position), in a bed without pillow, without blanket and without soft toy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France